CLINICAL TRIAL: NCT06285149
Title: Prospective Single-arm, Single-center Exploratory Clinical Study on Efficacy and Safety of Interventional Therapy Combined With Icaritin in First-line Treatment of Middle and Advanced HCC in Child Grade B Patients
Brief Title: Tace With Icaritin in First-line Treatment of Middle and Advanced HCC in Child Grade B Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKLD-22
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2023-12

CONDITIONS: HCC
MeSH Terms: interventions — icaritin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 80 patients with advanced HCC in Child-Pugh B who had not been systematically (Experimental): Icaritin will be divided into the first dose group (200mg bid orally) using 3+3 dosage. The second dose group will be 400mg bid orally; And the third dose group, 600mg bid, taken orally. It is taken within 1 hour after a meal, and Icaritin will be administered continuously during interventional therapy.
  Interventions: Drug: Icaritin

INTERVENTIONS:
Drug: Icaritin — This product is suitable for patients with unresectable hepatocellular carcinoma who are not suitable for or refuse to receive standard treatment and have not received systemic treatment in the past, and the peripheral blood compound markers of patients meet at least two of the following detection indicatorsItem: AFP>400 ng/mL; TNF-a<2.5 pg/mL; IFN-y>7.0 pg/mL.The conditional approval is based on data from an interim analysis of an enriched population in a randomized controlled Phase 11 clinical trial, and full approval for this indication will be subject to confirmation of the clinical benefit of the product in planned confirmatory trials.

SUMMARY:
Icaritin is a drug that has been approved by the National Medical Products Administration (NMPA) based on a multicenter, randomized, double-blind, parallel-controlled Phase III clinical trial - SNG1705 ICR-1. It is used for patients with unresectable hepatocellular carcinoma who are not suitable for or refuse standard treatment and have not previously received systemic therapy. According to numerous studies, in tumor cells, Icaritin can downregulate the expression of TNF-α, IL-6, PD-L1 and exert anti-tumor effects. At the same time, it regulates the tumor immune microenvironment by reducing the secretion of TNFa and IL-6 as well as inhibiting PD-L1 expression through decreasing MDSC cell proportion. Importantly, Icaritin has excellent safety profile and greatly ensure patients' quality of life clinically. Rare grade 3-4 TRAEs were observed in clinical trials which is uncommon among existing standard drugs. Good safety is a prerequisite for combination therapy; therefore, further exploration of optimal drug combinations is worth considering. Thus, TACE+Icaritin may potentially optimize treatment strategies for patients with poor liver function reserve.

DETAILED DESCRIPTION:
Child B patients have a lower tolerance to targeted immunotherapy, and combining interventional therapy with targeted immunotherapy can result in an accumulation of toxic side effects leading to disease progression. Additionally, repeated local interventions can further deteriorate liver function. These patients currently face limited treatment choices. Apatinib has minimal adverse reactions and has been recommended by experts as a level I option for Child B patients in the HCC 2022 CSCO guidelines. Therefore, combining interventional therapy with apatinib holds promise in improving survival outcomes for Child B patients.

ELIGIBILITY:
Inclusion Criteria:

1. HCC was confirmed by histopathology or clinical diagnosis;
2. No previous systematic therapy;
3. Age 18-75 years old;
4. CNLC: Ⅱb-Ⅲa stage;
5. Child-Pugh grade B;
6. ECOG PS score :0-1;
7. No major vessel invasion or distant metastasis;
8. Suitable for interventional treatment;
9. Measurable disease according to mRECIST;
10. Willing to sign informed consent;
11. Willing and able to follow study protocols and visit plans.

Exclusion Criteria:

1. Patients who refuse or are not suitable for interventional treatment;
2. Fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma and other components previously confirmed by histology/cytology;
3. Prior systematic therapy for HCC, including chemotherapy agents, sorafenib, Renvastinib, regorafenib and other targeted agents or immunomodulators such as anti-PD-1, anti-PD-L1, anti-CTLA-4, other than antiviral therapy for patients receiving any other investigational drug;
4. Contraindications for interventional therapy, such as severe cirrhosis, more than moderate ascites, and Child C liver function; 5, diagnosed as hepatic encephalopathy, sclerosing cholangitis, Gilbert disease;

6. A history of gastrointestinal bleeding or a definite tendency to gastrointestinal bleeding within the previous 6 months; 7. Serious dysfunction of vital organs such as heart, brain and lungs; 8.uncontrolled high blood pressure, gastrointestinal bleeding or coagulation dysfunction, etc.; 9. Pregnant or nursing patients; 10. Allergic to drugs or excipients used in the study; 11. Other conditions deemed inappropriate for participation in the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 years
  The proportion of patients with optimal response achieving complete or partial response
PFS | 2 years
  If the patient has not progressed or died at the last follow-up, the date on which the clinician last confirmed that there was no tumor progression will prevail. For patients who are lost to follow-up, the date when the tumor was last recorded as not progressing will be considered. Patients who have started a new treatment prior to progression will have the date their tumor was last recorded prior to the new treatment.

SECONDARY OUTCOMES:
Overall survival，OS | 2 years
  If the patient is still alive at the last follow-up, the date of the clinician's last confirmation of the patient's survival shall prevail. For patients who were lost to follow-up, the date of last recorded patient survival was considered.